CLINICAL TRIAL: NCT03167190
Title: Ultrasound-localized Landmark Identification in Hospitalized Patients Requiring Lumbar Puncture: Implications for Safety, Quality, and Procedural Success
Brief Title: Ultrasound-Assisted Lumbar Puncture
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Failed to meet target enrollment
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Michael P Boniface, M.D., Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 17-000511
Record Dates: First submitted 2017-05-24; First posted 2017-05-25 (Actual); Last update posted 2020-01-09 (Actual); Status verified 2020-01

CONDITIONS: Spinal Puncture; Diagnostic Imaging
Keywords: Point of Care Ultrasound

STUDY DESIGN:
Intervention Model Description: Participants will be enrolled into the control group (Landmark-based palpation and skin marking) vs the experimental group (ultrasound assisted identification of bony landmarks and skin marking).
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Other): Traditional landmark-based lumbar puncture technique by palpation
  Interventions: Procedure: Traditional Landmark-based Lumbar Puncture
- Experimental (ultrasound) (Experimental): Use of point-of-care ultrasound to identify bony landmarks.
  Interventions: Procedure: Point-of-care ultrasound

INTERVENTIONS:
Procedure: Point-of-care ultrasound — A point-of-care ultrasound machine will be utilized to identify and mark midline and the interspinous space based on visualization of spinous processes.
  Arms: Experimental (ultrasound)
Procedure: Traditional Landmark-based Lumbar Puncture — Palpation of anatomical landmarks to identify midline and interspinous space
  Arms: Control

SUMMARY:
Although the lumbar puncture is a common procedure and has been performed without ultrasound for decades, other research studies suggest that there may be some benefits to using ultrasound. This study intends to see whether by using ultrasound there is increased success rate, decreased need for additional procedures, and less discomfort during the procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who registered for an emergency or inpatient encounter between 5/22/2017 and 5/08/2018
2. Males or females 18 years of age or older
3. Patients who have been identified as requiring a lumbar puncture for any therapeutic or diagnostic or therapeutic indication, as decided by the neurology staff physicians, residents, or advanced practice providers.

Exclusion Criteria:

1. Patients who are not capable of providing consent for participation in research and do not have an authorized relative or power of attorney to consent in their stead.
2. Patients who require lumbar puncture in an emergency, time dependent fashion and in whom a possible delay could conceivable have a negative clinical impact.
3. Patients with known abnormal lumbar spinal anatomy or prior extensive surgical fusion such that fluoroscopic or CT guidance is determined to be more clinically appropriate by the treating physicians.
4. BMI greater than 60
5. Absolute contraindication to lumbar puncture such as uncorrected coagulopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2017-05-25 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Mean Procedural Duration | Approximately 1 hour
  This is defined by number of minutes from initiating of patient positioning (prior to evaluation of the anatomical landmarks) to first flow of cerebrospinal fluid (CSF).

SECONDARY OUTCOMES:
Number of Procedures Considered to be Failures | Approximately 1 hour
  As defined by inability to obtain cerebrospinal fluid despite multiple attempts, terminated at the discretion of the procedurist as would otherwise be clinically determined.
Number of Fluoroscopically Guided or CT Guided Lumbar Punctures | Approximately 7 days
  In the event of ultrasound procedural failure by clinician
Total number of unique skin punctures | Approximately 1 day
  This will be defined by the needle bevel completely exiting and skin and being re-inserted, during the duration of the procedure, whether the procedure is ultimately successful or not.
Procedurist reported ease of the procedure | Approximately 1 day
  Procedurist reported ease of the procedure will be reported by a 10 cm visual analog scale, with 0=easy and 10=very difficult.
Patient reported discomfort | Approximately 1 day
  Patient reported discomfort will be reported by a 10 cm visual analog scale, with 0=no discomfort and 10=extreme discomfort.
Number of red blood cells in collected CSF | Approximately 1 day
  This will be abstracted manually from the patient's electronic medical record.
Hospital Length of Stay | Approximately 1 month
  This will be abstracted manually from the patient's electronic medical record.

CONTACTS AND LOCATIONS:
Overall Officials: Michael P Boniface, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

REFERENCES:
- [Background] Edwards C, Leira EC, Gonzalez-Alegre P. Residency training: a failed lumbar puncture is more about obesity than lack of ability. Neurology. 2015 Mar 10;84(10):e69-72. doi: 10.1212/WNL.0000000000001335. PMID 25754807
- [Background] Engedal TS, Ording H, Vilholm OJ. Changing the needle for lumbar punctures: results from a prospective study. Clin Neurol Neurosurg. 2015 Mar;130:74-9. doi: 10.1016/j.clineuro.2014.12.020. Epub 2015 Jan 6. PMID 25590665
- [Background] Ferre RM, Sweeney TW. Emergency physicians can easily obtain ultrasound images of anatomical landmarks relevant to lumbar puncture. Am J Emerg Med. 2007 Mar;25(3):291-6. doi: 10.1016/j.ajem.2006.08.013. PMID 17349903
- [Background] Grau T, Leipold RW, Conradi R, Martin E, Motsch J. Ultrasound imaging facilitates localization of the epidural space during combined spinal and epidural anesthesia. Reg Anesth Pain Med. 2001 Jan-Feb;26(1):64-7. doi: 10.1053/rapm.2001.19633. No abstract available. PMID 11172514
- [Background] Huang MY, Lin AP, Chang WH. Ultrasound-assisted localization for lumbar puncture in the ED. Am J Emerg Med. 2008 Oct;26(8):955-7. doi: 10.1016/j.ajem.2008.03.007. No abstract available. PMID 18926360
- [Background] Lahham S, Schmalbach P, Wilson SP, Ludeman L, Subeh M, Chao J, Albadawi N, Mohammadi N, Fox JC. Prospective evaluation of point-of-care ultrasound for pre-procedure identification of landmarks versus traditional palpation for lumbar puncture. World J Emerg Med. 2016;7(3):173-7. doi: 10.5847/wjem.j.1920-8642.2016.03.002. PMID 27547275
- [Background] Nomura JT, Leech SJ, Shenbagamurthi S, Sierzenski PR, O'Connor RE, Bollinger M, Humphrey M, Gukhool JA. A randomized controlled trial of ultrasound-assisted lumbar puncture. J Ultrasound Med. 2007 Oct;26(10):1341-8. doi: 10.7863/jum.2007.26.10.1341. PMID 17901137
- [Background] Peterson MA, Pisupati D, Heyming TW, Abele JA, Lewis RJ. Ultrasound for routine lumbar puncture. Acad Emerg Med. 2014 Feb;21(2):130-6. doi: 10.1111/acem.12305. PMID 24673668
- [Background] Williams S, Khalil M, Weerasinghe A, Sharma A, Davey R. How to do it: bedside ultrasound to assist lumbar puncture. Pract Neurol. 2017 Jan;17(1):47-50. doi: 10.1136/practneurol-2016-001463. Epub 2016 Nov 28. PMID 27895189
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials